CLINICAL TRIAL: NCT05829928
Title: Testicular Tissue Cryopreservation in the Setting of Gender-Affirming Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: STUDY19070264
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria; Transgender
Keywords: Fertility; Fertility Preservation; Infertility; Gender Affirming; Gender Diverse; Non-Binary
MeSH Terms: conditions — Gender Dysphoria; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Testicular Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cryopreservation: Participants will have gonadal tissue removed and cryopreserved for future fertility applications.
  Interventions: Diagnostic Test: Infectious Disease Testing; Procedure: Gonadal Tissue Removal

INTERVENTIONS:
Diagnostic Test: Infectious Disease Testing — Participants will undergo infectious disease testing.
Procedure: Gonadal Tissue Removal — Removal of gonadal tissue will be done through a surgical procedure.

SUMMARY:
The goal of this study is to learn about fertility preservation in the gender-diverse community. The main objectives it aims to understand are to:

1. Optimize techniques for processing and cryopreserving testicular tissue.
2. Determine presence and number of germ cells (sperm precursors) in the patients' testicular tissue.
3. Develop next generation cell- and tissue-based therapies for preserving fertility and treating infertility.

DETAILED DESCRIPTION:
Fertility preservation is an important aspect of care for all patients who may have their fertility compromised secondary to disease, medical treatments, age or other circumstances, including treatments for gender dysphoria. An increasing number of gender diverse patients are presenting to fertility clinics for fertility preservation. Studies indicate that parenthood is important for this patient population. Therefore, both the Endocrine Society and the World Professional Association for Transgender Health (WPATH) recommend that fertility preservation be discussed with all patients prior to initiation of medical treatments for gender dysphoria.

For gender diverse patients, medical treatment is primarily comprised of estradiol, which is often preceded by GnRH agonists (such as leuprolide acetate, histrelin) to reduce endogenous testosterone production. There are theoretical concerns about the effects of long-standing hormonal treatment on the gonads and future fertility potential. Regardless of the timing of initiation of hormone suppression and/or estradiol therapy, fertility preservation counseling is an essential aspect of their care. Sperm preservation does require the individual to undergo their natal puberty, and for many transgender patients, this is undesirable and even contra-indicated from mental health standpoint, as the suicide rate for transgender youth is 10-times the national average. Testicular tissue cryopreservation is an alternative option for transgender patients who desire pubertal blockade and estradiol but have not yet initiated sperm production (spermarche) to preserve their fertility. Spermarche typically occurs at sexual maturity rating (SMR) 4 and pubertal blockade is offered as early as SMR 2.

ELIGIBILITY:
Inclusion Criteria:

Category 1 participants must have all criteria listed below:

* Patient with testes over the age of 9
* Diagnosed with gender dysphoria; currently on or imminently planning to start gender affirming treatment (hormone blockers or gender-affirming hormones)
* Have a clinical referral for fertility preservation from their primary care physician
* Unwilling to undergo natal puberty or, for patients who have gone through puberty, unwilling to discontinue hormone suppression and/or hormone replacement therapy.

Category 2 participants only fall into this category if they are undergoing gender-affirming surgery. They must have all criteria listed below:

* Patient is 18+ years old
* Diagnosed with gender dysphoria
* Unwilling to undergo natal puberty, or for patients who have gone through puberty, be unwilling to discontinue hormone suppression and/or sex steroid (estrogen) therapy.
* Will be undergoing gender affirming surgery that involves removal of the testes.

Exclusion Criteria:

* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Min Age: 9 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients who will undergo gender-affirming treatments and for whom standard of care fertility preservation procedures are not available.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Optimization of testicular tissue/cell cryopreservation techniques | [10 years]
  Testicular tissue will be used to isolate a suspension of testicular cells using a series of enzymatic digestions, washes, and filtrations. Testicular cells donated to the research pool will be frozen using varying cryopreservation methods and thawed to determine the efficacy of the freeze/thaw techniques. The concentration and number of recovered spermatogonial stem cells in the thawed cells will be determined using a human-to-nude mouse xenotransplantation assay. Recovery of spermatogonial stem cells will be compared to the concentration and number prior to cryopreservation using the same assay. Data gathered from this research will assist in identifying and overcoming some of the challenges to successful freezing and thawing of cells for future use by the patient.
To determine presence and number of germ cells (sperm precursors) in the patients' testicular tissue | [10 years]
  The number of stem cells in the developing testis in the humans is currently not established. Therefore, a small piece of testicular tissue from each patient (from the research portion) will be fixed in 4% of paraformaldehyde (PFA) and stained for known germ cell markers in order to count the number of stem cells in the patient tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/ University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish individual participant data. The investigators will also report each individual participant's data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: We will share IPD with the patients (and only the patient) within one year of enrollment. We share study protocol and ICF with collaborating sites upon request. De-identified IDP is shared with collaborating sites annually.
Access Criteria: De-identified research data will be shared with collaborators via e-mail, and with the broader scientific community via publication and presentations at national/international meetings.